CLINICAL TRIAL: NCT03086447
Title: Evaluation of Astigmatic Contact Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR-5871
Record Dates: First submitted 2017-03-16; First posted 2017-03-22 (Actual); Results first posted 2018-07-10 (Actual); Last update posted 2018-07-10 (Actual); Status verified 2018-06

CONDITIONS: Visual Acuity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Experimental: Participating Subjects (Experimental): Subjects who are habitual soft toric contact lens wearers, aged 18 to 40 years of age, will be dispensed the investigational contact lens to be worn from 28-36 days, to include a total of 5 visits.
  Interventions: Device: Investigational Contact Lens
- Control: Participating Subjects (Active Comparator): Subjects who are habitual soft toric contact lens wearers, aged 18 to 40 years of age, will be dispensed marketed contact lens to be worn from 28-36 days, to include a total of 5 visits.
  Interventions: Device: Marketed Contact Lens

INTERVENTIONS:
Device: Investigational Contact Lens — Senofilcon C Toric
  Arms: Experimental: Participating Subjects
Device: Marketed Contact Lens — Air Optix for Astigmatism
  Arms: Control: Participating Subjects

SUMMARY:
Randomized, double-masked, 5-visit, bilateral dispensing, parallel group study to demonstrate that the investigational contact lens meets the design requirements related to corneal staining, lens fit, visual acuity and rotational performance as well as subjective comfort and handling. Subjects will wear the contact lenses for a total of 28-36 days.

ELIGIBILITY:
Inclusion Criteria:

* 1) Healthy adult males or females age ≥18-40 years of age with signed informed consent.

  2) The subject must appear able and willing to adhere to the instructions set forth in this clinical protocol.

  3) Subject must be a habitual soft toric contact lens wearer. Habitual wearer is defined as someone who wears contact lenses for at least 6 hours a day, 5 days a week for the past 30 days.

  4) Subject's vertex corrected spherical component of their distance refraction must be between -1.00 to -4.75 Diopter (D) (inclusive) in each eye.

  5) Subject's vertex corrected refractive cylinder must be between -0.75 and -1.50 DC (inclusive) in each eye.

  6) Subject's refractive cylinder axis must be 180±25 and 90±15 in each eye. 7) The subject must have visual acuity best correctable to 20/25 or better for each eye 8) The subject must read and sign the Informed Consent form.

Exclusion Criteria:

* 1) Women who are pregnant or breastfeeding, 2) Any ocular or systemic allergies or diseases that may contraindicate contact lens wear.

  3) Any ocular medications use within the last one month. 4) Any systemic disease, autoimmune disease, or use of medication, which may interfere with contact lens wear.

  5) Any infectious disease (e.g., hepatitis, tuberculosis) or a contagious immunosuppressive disease (e.g., HIV), by self-report.

  6) Habitual wearer of extended wear contact lenses. 7) Known sensitivity to Revitalens OcuTec® 8) Any previous history of ocular and/or refractive surgery (e.g., radial keratotomy, PRK, LASIK, etc.).

  9) A clinical finding or history of entropion, ectropion, extrusions, chalazia, recurrent styes, glaucoma, history of recurrent corneal erosions, aphakia, or moderate or above corneal distortion, by self-report.

  10) History of binocular vision abnormality or strabismus, by self-report. 11) Habitual wearer of rigid gas permeable (RGP) lenses, orthokeratology lenses, or hybrid lenses (e.g. SynergEyes, SoftPerm) within the past 6 months.

  12) Employee of investigational clinic (e.g., Investigator, Coordinator, Technician).

  13) Participation in any contact lens or lens care product clinical trial within 14 days prior to study enrollment.

  14) Clinically significant (grade 3 or higher) corneal edema, corneal vascularization, corneal staining, tarsal abnormalities, bulbar injection or any other abnormalities which would contraindicate contact lens wear.

  15) Any history of a contact lens-related corneal inflammatory event within the past year that may contraindicate contact lens wear.

  16) Any active ocular infection. 17) Any corneal distortion resulting from previous hard or rigid gas permeable contact lens wear.

  18) Any fluctuations in vision due to clinically significant dry eye or other ocular conditions.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 267 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2017-05-04 (Actual); Study Completion 2017-05-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (17):
- United States (17):
  - Golden Optometric Group, Whittier, California
  - Dr. James Weber & Associates, PA, Jacksonville, Florida
  - Edward S. Wygonik, OD, Jacksonville Beach, Florida
  - Sabal Eye Care, Longwood, Florida
  - Maitland Vision Center, Maitland, Florida
  - Indiana University School of Optometry, Bloomington, Indiana
  - Kannarr Eye Care, Pittsburg, Kansas
  - ABQ Eye Care, Albuquerque, New Mexico
  - Sacco Eye Group, Vestal, New York
  - ProCare Vision Centers, Granville, Ohio
  - EyeCare Professionals of Powell, Powell, Ohio
  - Professional Vision Care, Inc, Westerville, Ohio
  - West Bay Eye Associates, Warwick, Rhode Island
  - Total Eye Care, PA, Memphis, Tennessee
  - Premier Vision, Amarillo, Texas
  - William J Bogus, OD, FAAO, Salt Lake City, Utah
  - Botetourt Eyecare, LLC, Salem, Virginia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 267 subjects were enrolled into this study. Of the enrolled 262 were randomized to receive a study lens, while 5 subjects failed to meet the eligibility criteria. Of the 262 randomized subjects, 231 completed the study and 31 subjects were discontinued.
Pre-assignment Details: One subject was randomized to the Test lens but in actuality was dispensed the control lens, therefore his/her data was summarized with the control data, while this/her demographic information is apart of the Test summary.
Groups:
- Lotrafilcon B (Control): Subjects that wore the lotrafilcon B lens throughout the entire duration of the study.
- Senofilcon C Toric (Test): Subjects that wore the senofilcon C toric lens throughout the entire duration of the study.
Period: Overall Study
Arm/Group | Lotrafilcon B (Control) | Senofilcon C Toric (Test)
Started | 132 | 130
Completed | 121 | 110
Not Completed | 11 | 20
Not completed — No Longer Meets Eligibility Criteria | 0 | 1
Not completed — Lost Lens | 2 | 5
Not completed — Product quality complaint | 0 | 1
Not completed — Lens Damage | 1 | 6
Not completed — Unsatisfactory Lens Fitting | 0 | 1
Not completed — Test Article No Longer Available | 1 | 0
Not completed — Protocol Violation | 2 | 4
Not completed — Lost to Follow-up | 0 | 1
Not completed — Adverse Event | 3 | 0
Not completed — Lens Discomfort | 2 | 1

BASELINE CHARACTERISTICS:
Population: All subjects that were randomized to a study lens.
Groups:
- Total: Total of all reporting groups
Arm/Group | Lotrafilcon B (Control) | Senofilcon C Toric (Test) | Total
Number analyzed (Participants) | 132 | 130 | 262
Age, Continuous [Mean (Standard Deviation); unit: Years] | 29.3 (6.50) | 29.4 (5.81) | 29.4 (6.16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 95 | 74 | 169
  Male | 37 | 56 | 93
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 2
  Asian | 6 | 4 | 10
  Black or African American | 13 | 12 | 25
  Native Hawaiian or Other Pacific | 1 | 0 | 1
  White | 110 | 111 | 221
  Other | 2 | 1 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 132 | 130 | 262

OUTCOME MEASURES:

1. Primary Outcome: Monocular Distance Visual Acuity (VA)
Description: Monocular distance visual acuity was measured with the study lens using a Snellen distance VA chart at an optical distance of 20 feet throughout the study. Observed VA data collected during all planned visits were dichotomized whether VA was "20/40 or better (acceptable VA)" or "worse than 20/40 (unacceptable VA)". VA of 20/40 with a negative modifier was considered worse than 20/40. The number of eye with acceptable VA was reported for each study lens.
Time Frame: Up to 4-Week Follow-up
Population: All subjects who administered the test article and have at least one observation after lens insertion.
Measure: Number; unit: Eyes
Units Other Than Participants: Number of Eyes
Arm/Group | Senofilcon C Toric (Test) | Lotrafilcon B (Control)
Number analyzed (Participants) | 129 | 132
Number analyzed (Number of Eyes) | 258 | 264
Eyes | 258 | 263
Statistical Analysis 1: Comparison: Senofilcon C Toric (Test); Proportion of eyes with overall acceptable VA assessed throughout the study period (up to 4-week) in the Test group was compared to the historical control acceptable rate of 80%. Lower 95% confidence limit was compared to 0.8; Test type: Other — It was deemed that a total of 135 subjects in the Test group is sufficient to demonstrate statistical acceptance of monocular VA better than equal to 20/40 with a minimum of 90% statistical power using the reference incidence rate of 95% with a correlation of 0.8 between eyes; Binomial proportion with Agresti-Coull — All primary hypotheses were simultaneously evaluated using a significance level of 0.05 following the intersection-union principal. All primary hypotheses must be met to claim success of the study objectives; Proportion = 100, 95% CI 2-sided [96.5 to 100] — All eyes (100%) in the Test group had acceptable VA throughout the study

2. Primary Outcome: Lens Fit Acceptance
Description: Lens fit characteristics were assessed using slit lamp with respect to lens position, movement and tightness. Each lens fit collected at fitting (visit 1) was judged being either acceptable or unacceptable based on the static and dynamic fit characteristic. The number of eyes with acceptable lens fit was reported for each study lens.
Time Frame: 15 Minutes Post Lens Fitting
Population: All subjects who administered the test article and have at least one observation after lens insertion.
Measure: Number; unit: Eyes
Units Other Than Participants: Number of Eyes
Arm/Group | Senofilcon C Toric (Test) | Lotrafilcon B (Control)
Number analyzed (Participants) | 129 | 132
Number analyzed (Number of Eyes) | 258 | 264
Eyes | 258 | 264
Statistical Analysis 1: Comparison: Senofilcon C Toric (Test); Proportion of eyes with acceptable lens fit assessed at fitting (visit 1) in the Test group was compared to the historical control rate of 80%. Lower 95% confidence limit was compared to 0.8; Test type: Other — It was deemed that a total of 135 subjects in the Test group is sufficient to demonstrate statistical acceptance of lens fit with a minimum of 90% statistical power using the reference incidence rate of 95% with a correlation of 0.8 between eyes; Binomial proportion with Agrestic-Coull — [p-value comment as in outcome 1, analysis 1]; Proportion = 100.0, 95% CI 2-sided [96.5 to 100.0] — All eyes (100%) in the Test group had acceptable lens fit at fitting (visit 1)

3. Primary Outcome: Lens Stability With Blink
Description: Lens rotational stability with blink was assessed using slit lamp with beam that can be rotated. The stability of the scribe mark rotational position during a series of normal (unforced) blinks was assessed, and then dichotomized whether stability was less than or equal to 5-degree (acceptable stability) or greater (unacceptable stability). The number of eye with acceptable stability was reported for each lens.
Time Frame: 15 Minutes Post Lens Fitting
Population: All subjects who administered the test article and have at least one observation after lens insertion.
Measure: Number; unit: Eyes
Units Other Than Participants: Number of Eyes
Arm/Group | Senofilcon C Toric (Test) | Lotrafilcon B (Control)
Number analyzed (Participants) | 129 | 132
Number analyzed (Number of Eyes) | 258 | 264
Eyes | 258 | 264
Statistical Analysis 1: Comparison: Senofilcon C Toric (Test); Proportion of eyes with acceptable stability assessed at fitting (visit 1) in the Test group was compared to the historical control rate of 80%. Lower 95% confidence limit was compared to 0.8; Test type: Other — It was deemed that a total of 135 subjects in the Test group is sufficient to demonstrate statistical acceptance of lens stability with a minimum of 90% statistical power using the reference incidence rate of 95% with a correlation of 0.8 between eyes; Binomial proportion with Agrestic-Coull — [p-value comment as in outcome 1, analysis 1]; Proportion = 100.0, 95% CI 2-sided [96.5 to 100.0] — All eyes (100%) in the Test group had acceptable stability at fitting

4. Primary Outcome: Absolute Lens Rotation
Description: Lens rotation was assessed using slit lamp with beam that can be rotated. The rotational error (assume shortest distance) and direction (base toward the nose or temple) were calculated, and then absolute rotation was dichotomized whether absolute rotation was less than or equal to 10-degree (acceptable rotation) or greater (unacceptable rotation). The number of eyes with acceptable lens rotation for each lens was reported.
Time Frame: 15-minutes Post Lens Insertion
Population: All subjects who administered the test article and have at least one observation after lens insertion.
Measure: Number; unit: Eyes
Units Other Than Participants: Number of Eyes
Arm/Group | Senofilcon C Toric (Test) | Lotrafilcon B (Control)
Number analyzed (Participants) | 129 | 133
Number analyzed (Number of Eyes) | 258 | 266
Eyes | 255 | 261
Statistical Analysis 1: Comparison: Senofilcon C Toric (Test); Proportion of eyes with acceptable absolute rotation assessed at 15-minute upon insertion (fitting, visit 1) in the Test group was compared to the historical control rate of 80%. Lower 95% confidence limit was compared to 0.8; Test type: Other — It was deemed that a total of 135 subjects in the Test group is sufficient to demonstrate statistical acceptance of absolute rotation with a minimum of 90% statistical power using the reference incidence rate of 95% with a correlation of 0.8 between eyes; Linear mixed model with binomial dist. — [p-value comment as in outcome 1, analysis 1]; Least square mean proportion = 99.6, 95% CI 2-sided [97.5 to 99.9] — Above 80% of eyes in the Test group had acceptable rotation

5. Primary Outcome: Corneal Staining
Description: Contact lens related corneal staining was assessed using slit lamp throughout the study. Corneal staining was graded using a 5-level scale: 0=no staining, 1=trace, 2=mild, 3=moderate and 4=severe. Corneal staining data collected during planned and unplanned visits were dichotomized whether the level of corneal stating was grade 3 or higher (unacceptable CS) or less than grade 3 (acceptable CS). The number of eyes with Grade 3 or higher was reported for each lens type.
Time Frame: Up to 4-Week Follow-up
Population: All subjects who administered the test article and have at least one observation after lens insertion.
Measure: Number; unit: Eyes
Units Other Than Participants: Number of Eyes
Arm/Group | Senofilcon C Toric (Test) | Lotrafilcon B (Control)
Number analyzed (Participants) | 129 | 133
Number analyzed (Number of Eyes) | 258 | 266
Eyes | 0 | 3
Statistical Analysis 1: Comparison: Senofilcon C Toric (Test) vs Lotrafilcon B (Control); Proportion of eyes with unacceptable corneal staining (CS) throughout all planned and unplanned visits in the Test group was compared to that in the Control group; Test type: Other — It was deemed that a total of 135 subjects per each study group is sufficient to demonstrate no statistical difference in the CS incidence rate between the Test and Control groups with a minimum of 80% statistical power using the reference incidence rate of 0.005% with a correlation of 0.3 between eyes within subject; Bayesian beta-binomial model — [p-value comment as in outcome 1, analysis 1]; A 95% credible interval for the posterior estimate (Test over Control) was used to test no difference between the Test and Control groups; Odds Ratio (OR) = 0.29, 95% CI 2-sided [0.004 to 1.437] — odds ratio calculated as Test over Control

6. Secondary Outcome: Overall Comfort
Description: Overall comfort was assessed using the Contact Lens User Experience™ (CLUE) questionnaire. CLUE is a validated patient-reported outcomes (PRO) questionnaire to assess patient-experience attributes of soft contact lenses (comfort, vision, handling, and packaging) in a contact-lens wearing population in the US, ages 18-65. Derived CLUE scores using Item Response Theory (IRT) follow a normal distribution with a population average score of 60 (SD 20), where higher scores indicate a more favorable/positive response with a range of 0-120.
Time Frame: Up to 4- Week Follow-up
Population: All subjects who have successfully completed all required visits without any major protocol deviations.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Senofilcon C Toric (Test) | Lotrafilcon B (Control)
Number analyzed (Participants) | 108 | 120
Units on a Scale | 61.4 (23.45) | 52.0 (24.45)
Statistical Analysis 1: Comparison: Senofilcon C Toric (Test) vs Lotrafilcon B (Control); Sample size calculation was performed considering the effect size of 5 (Test minus Control) to achieve a minimum statistical power of 90% at a 5% significance level; Test type: Non-Inferiority — A non-inferiority margin of -5 points was used. This margin is based on a 10% shift in the distribution of CLUE score; Linear mixed model; A 95% confidence interval for the least square mean difference was used to demonstrate non-inferiority of the Test relative to the Control groups; Mean Difference (Final Values) = 6.8, 95% CI 2-sided [2.1 to 11.5], Standard Deviation 2.39 — Mean difference was calculated as Test minus Control

7. Secondary Outcome: Overall Handling
Description: Overall Handling was assessed using the Contact Lens User Experience™ (CLUE) questionnaire. CLUE is a validated patient-reported outcomes (PRO) questionnaire to assess patient-experience attributes of soft contact lenses (comfort, vision, handling, and packaging) in a contact-lens wearing population in the US, ages 18-65. Derived CLUE scores using Item Response Theory (IRT) follow a normal distribution with a population average score of 60 (SD 20), where higher scores indicate a more favorable/positive response with a range of 0-120.
Time Frame: Up to 4- Week Follow-up
Population: All subjects who have successfully completed all required visits without any major protocol deviations.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Senofilcon C Toric (Test) | Lotrafilcon B (Control)
Number analyzed (Participants) | 108 | 120
Units on a Scale | 63.5 (20.90) | 65.7 (19.77)
Statistical Analysis 1: Comparison: Senofilcon C Toric (Test) vs Lotrafilcon B (Control); [analysis description as in outcome 6, analysis 1]; Test type: Non-Inferiority — A non-inferiority margin of -5 points was used. This margin is based on a 10% shift in the distribution of CLUE score; Linear mixed model; [statistical method as in outcome 6, analysis 1]; Mean Difference (Final Values) = -3.1, 95% CI 2-sided [-7.2 to 0.9], Standard Deviation 2.04 — Mean difference was calculated as Test minus Control

8. Secondary Outcome: Monocular Distance Visual Acuity (VA)
Description: Monocular distance visual acuity was measured with the study lens using a Snellen distance VA chart at an optical distance of 20 feet. Observed VA data collected at fitting were dichotomized whether VA was "20/20 or better (optimal VA)" or "worse than 20/20". VA of 20/20 with a negative modifier was considered worse than 20/20. The number of eyes with 20/20 vision was reported for each study lens.
Time Frame: 15 Minutes Post Lens Fitting
Population: All subjects who have successfully completed all required visits without any major protocol deviations.
Measure: Number; unit: Eyes
Units Other Than Participants: Number of Eyes
Arm/Group | Senofilcon C Toric (Test) | Lotrafilcon B (Control)
Number analyzed (Participants) | 108 | 120
Number analyzed (Number of Eyes) | 216 | 240
Eyes | 177 | 184
Statistical Analysis 1: Comparison: Senofilcon C Toric (Test); Proportion of eyes with optimal VA assessed at fitting in the Test group was compared to the Control group; Test type: Non-Inferiority — A non-inferiority margin of 0.5 was used. This margin is based on a 10% difference in the distribution between the Test and Control groups; Generalized LMM w/ binomial dist; Odds Ratio (OR) = 1.77, 95% CI 2-sided [0.98 to 3.22] — Odds ratio of Test over Control was calculated

ADVERSE EVENTS:
Time Frame: Throughout the duration of the study. Approximately 1 month per subject.
Arm/Group | Lotrafilcon B (Control) | Senofilcon C Toric (Test)
All-Cause Mortality (participants affected / at risk) | 0/132 | 0/130
Serious Adverse Events (participants affected / at risk) | 0/132 | 0/130
Other Adverse Events (participants affected / at risk) | 0/132 | 0/130

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2017-03-14): https://cdn.clinicaltrials.gov/large-docs/47/NCT03086447/Prot_000.pdf
  • Statistical Analysis Plan (2017-05-22): https://cdn.clinicaltrials.gov/large-docs/47/NCT03086447/SAP_001.pdf